

# **Study Information**

| Title | Compare Effectiveness of Tofacitinib 11 mg |
|---|---|
| | QD to Tofacitinib 5 mg BID |
| Protocol number | A3921359 |
| Protocol version identifier | 1.0 |
| Date | 10 December 2019 |
| Active substance | Tofacitinib citrate |
| Medicinal product | Xeljanz (tofacitinib) |
| Research question and objectives | Main objective is to compare effectiveness of tofacitinib 11 mg once daily (QD) initiators to tofacitinib 5 mg twice daily (BID) initiators |
| Author | PPD PPD PPD PPD PPD PPD |

# 1. TABLE OF CONTENTS 2. LIST OF ABBREVIATIONS......4 5. AMENDMENTS AND UPDATES......7 6. MILESTONES ......8 7. RATIONALE AND BACKGROUND......8 8. RESEARCH QUESTION AND OBJECTIVES ......9 9. RESEARCH METHODS ......9 10. PROTECTION OF HUMAN SUBJECTS ......14 10.3. Institutional Review Board (IRB)/Independent Ethics Committee (IEC) ......14 11. MANAGEMENT AND REPORTING OF ADVERSE EVENTS/ADVERSE REACTIONS .......14 12. PLANS FOR DISSEMINATING AND COMMUNICATING STUDY RESULTS.......14

# Tofacitinib A3921359 NON-INTERVENTIONAL STUDY PROTOCOL Final V1.0, 10 December 2019

| 14. LIST OF TABLES | 16 |
|-----------------------------------------------|----|
| 15. LIST OF FIGURES | 16 |
| ANNEX 1. LIST OF STAND ALONE DOCUMENTS | 16 |
| ANNEX 2. ENCEPP CHECKLIST FOR STUDY PROTOCOLS | 16 |
| ANNEX 3. ADDITIONAL INFORMATION | 16 |

# 2. LIST OF ABBREVIATIONS

| Abbreviation | Definition |
|--------------|----------------------------------------------------|
| ACR | American College of Rheumatology |
| AE | Adverse Event |
| BID | Twice daily |
| CDAI | Clinical Disease activity index |
| CRP | C- reactive protein |
| csDMARD | Conventional Disease modifying anti-rheumatic drug |
| DAS | Disease activity score |
| mDAS | Modified Disease Activity Score |
| EMA | European Medicines Agency |
| ESR | Erythrocyte sedimentation rate |
| EQ-5D | Euro Qol 5D |
| FDA | Food and Drug Administration |
| GPP | Good Pharmacoepidemiology Practices |
| GEP | Good Epidemiology Practices |
| mHAQ | modified Health Assessment questionnaire |
| HAQ | Health Assessment questionnaire |
| IEA | International Epidemiology Association |
| IEC | Independent Ethics Committee |
| IR | Immediate Release |
| IRB | Institutional Review Board |
| ISPE | International Society of Pharmacoepidemiology |
| JAK | Janus kinase |
| LDA | Low Disease Activity |
| LTE | Long Term Extension |
| MCID | Minimally clinically important difference |
| MR | Modified release |
| MTX | methotrexate |
| NI | Non Interventional |
| PD | Pharmacodynamic |
| PK | Pharmacokinetic |
| PS | Propensity Score |
| QD | Once daily |
| RA | Rheumatoid arthritis |
| SAP | Statistical analysis plan |
| SAS | Statistical Analysis System |
| TyK2 | Tyrosine kinase 2 |
| US | United States |

# 3. RESPONSIBLE PARTIES

| Name, degree(s) | Job Title | Affiliation | Address |
|-----------------|------------------------|--------------|---------|
| PPD MD | Global Medical Affairs | Pfizer, Inc. | PPD |
| | | | Spain |
| PPD PhD, | Epidemiologist – | Pfizer, Inc. | PPD |
| MPH | Non-Interventional | | |
| | Study lead | | USA |
| PPD | PPD | Corrona, LLC | ארט |
| MD, MPH | | | |
| | _ | | USA |
| PPD | PPD | Corrona, LLC | PPD |
| PhD | | | |
| | | | USA |

# 4. ABSTRACT

Not Applicable.

# 5. AMENDMENTS AND UPDATES

None.

#### 6. MILESTONES

| Milestone | Planned date |
|-----------------------------------|-------------------|
| Final approved protocol* | December 2019 |
| Start of analysis/data collection | 30 September 2018 |
| Approved SAP | 20 March 2018 |
| End of data collection | 30 August 2019 |
| Final study report | 11 October 2019 |

<sup>\*</sup> This protocol was created retrospective from start of data collection and is part of an Significant Qulaity Event (SQE).

#### 7. RATIONALE AND BACKGROUND.

Tofacitinib is a potent, selective inhibitor of the Janus kinase (JAK) family of kinases with a high degree of selectivity against other kinases in the human genome. In kinase assays, tofacitinib, inhibits JAK1, JAK2, JAK3, and to a lesser extent tyrosine kinase 2 (TyK2). In cellular settings where JAK kinases signal in pairs, tofacitinib preferentially inhibits signaling by heterodimeric receptors associated with JAK3 and/or JAK1 with functional selectivity over receptors that signal via pairs of JAK2. The efficacy and safety of tofacitinib 5 mg twice daily (BID) administered as monotherapy or in combination with conventional disease modifying anti rheumatic drugs (csDMARDs), mainly methotrexate (MTX), in patients with moderately to severely active rheumatoid arthritis (RA), have been demonstrated in Phase 2,<sup>1-5</sup> Phase 3,<sup>6-11</sup> and Phase 3b/4<sup>12</sup> studies of up to 24 months' duration, and in long-term extension (LTE) studies with up to 9.5 years of observation. <sup>13-15</sup>

The immediate release (IR) formulation of tofacitinib was approved in November 2012 in the US for the treatment of moderate to severe rheumatoid arthritis (RA) as a twice daily (BID) regimen. It was followed by Food and Drug Administration (FDA) approval of 11 mg modified release once daily (QD) dose in February of 2016.

The modified release (MR) QD regimen has the potential to improve drug compliance of patients, patient convenience, and to offer additional dosing options for patients. Data from completed pharmacokinetic (PK) studies demonstrated that the desired pharmacokinetic and pharmacodynamic (PK-PD) profile was achieved by the MR dose. Overall similarity of PK parameters between IR and MR formulations were found Phase 1 PK studies comparing MR and IR formulations. Therefore, based on the pharmacokinetic (PK) profile for the 2 formulations (IR and MR) and from the information obtained from IR BID programs, FDA approved MR based on clinical pharmacology studies.

It is hypothesized that patients prescribed to facitinib 11 mg MR formulation once daily (QD) will achieve similar benefit to those prescribed to facitinib 5 mg BID dosage in real world use. This study will therefore seek to compare the effectiveness of the MR 11 mg QD regimen to the IR 5 mg BID regimen for the treatment of RA in a real-world registry of RA patients.

## 8. RESEARCH QUESTION AND OBJECTIVES

# **Primary Objective:**

The overall aim of this study is to the compare clinical effectiveness of tofacitinib in patients initiating tofacitinib 11 mg QD or 5 mg BID identified from the Corrona US RA Registry.

# **Secondary Objective:**

The study also aims to descriptively assess effectiveness in patients that switched from tofacitinib 5 mg BID to tofacitinib 11 mg QD after February 2016.

#### 9. RESEARCH METHODS

### 9.1. Study Design

This is an observational study conducted in a cohort of tofacitinib-exposed patients to evaluate effectiveness of tofacitinib MR 11 mg QD tablet compared to IR 5 mg BID tablet. In this secondary data collection study of structured data, patient therapeutic strategies are not determined by this protocol.

# 9.2. Setting

Using the United States (US) Corrona RA Registry database, <sup>16</sup> patients with RA who have been exposed to tofacitinib IR or MR on or after February 2016 will be included in this study. In order to adequately measure the outcome, the initiators will also be required to have a follow-up visit at 6 months (+/- 3 months) after tofacitinib initiation.

For the primary analysis comparing QD to BID patients, we will consider those patients who initiated tofacitinib 5 mg BID on or after February 2016 and those that initiated tofacitinib 11 mg QD after it became available in February 2016. Although the sample size will be smaller than if all tofacitinib 5 mg BID patients were considered, the inclusion of those patients may introduce noise since there is the possibility that they could differ from the more recent initiators. Therefore, we will consider the cleaner cohort of all patients initiating tofacitinib on or after February 2016.

For the secondary aim, patients that switched from tofacitinib 5 mg BID to tofacitinib 11 mg QD ("switchers") will be considered. Patients will be considered to have switched from 5 mg BID to 11 mg QD if they initiated 5 mg BID after February 2016 and subsequently changed their dose to 11 mg QD.

# 9.2.1. Inclusion Criteria

Patients must meet all of the following inclusion criteria to be eligible for inclusion in the study:

1. All US Corrona RA Registry patients who initiated to facitinib 5 mg BID or to facitinib 11 mg QD after it became available in February 2016.

- 2. Patients must have a follow-up visit at 6 months (+/- 3 months) after tofacitinib initiation. These 6 month visits are part of routine practice and is not associated with this protocol.
- 3. Patients must have a valid clinical disease activity index (CDAI) at initiation and at 6-month follow-up visit.

#### 9.2.2. Exclusion Criteria

There are no exclusion criteria for this study.

#### 9.3. Variables

The US Corrona RA Registry is an efficient data collection system for evaluating a range of efficacy outcomes associated with therapies used to treat RA. The endpoints chosen for this study will be extracted from patient and physician questionnaires. Demographic data collected includes age, gender, race and ethnicity. In addition, baseline disease characteristics like disease duration and severity etc. will be captured for both the IR and MR cohorts under study to evaluate disease characteristics.

**Primary outcome**: Minimally clinically important difference (MCID) improvement as defined by difference in Clinical Disease activity index (CDAI) from initiation to 6 month visit. MCID is dependent on baseline disease activity (at initiation); MCID≥2 if CDAI at initiation of Low CDAI ≤10, MCID≥6 if CDAI at initiation Moderate of 10<CDAI≤22 and MCID≥11 if CDAI at initiation high of >22.

## **Secondary Outcomes:**

- Change in CDAI from baseline to 6 month follow-up (as a continuous variable).
- Achievement of Remission (CDAI\le 2.8) at 6 month follow-up (among all).
- Achievement of Remission (CDAI\le 2.8) at 6 month follow-up (among those that were not in remission at initiation).
- Achievement of Low Disease Activity (LDA) (CDAI≤10) at 6 month follow-up (among all).
- Achievement of Low Disease Activity (LDA) (CDAI≤10) at 6 month follow-up (among those that were not in remission or LDA at initiation).
- Achievement of improvement from baseline to 6 month follow-up in modified Health Assessment Questionnaire (mHAQ) of at least 0.25 (as a dichotomous variable).
- Achievement of improvement from baseline to 6 month follow-up in Health assessment questionnaire (HAQ) of at least 0.22.

- Change from baseline to 6 month follow-up HAQ (HAQ as a dichotomous variable).
- Change from baseline to 6 month follow-up modified HAQ (mHAQ as a continuous variable).
- Change from baseline to 6 month follow-up HAQ (HAQ as a continuous variable).
- Change from baseline to 6 month follow-up modified Disease activity Score (mDAS as a continuous variable).
- Change from baseline to 6 month follow-up Disease activity score- erythrocyte sedimentation rate (DAS ESR) (as a continuous variable).
- Change from baseline to 6 month follow-up DAS- C- reactive protein (DAS CRP) (as a continuous variable).
- Change from baseline to 6 month follow-up patient pain (as a continuous variable).
- Change from baseline to 6 month follow-up patient fatigue (as a continuous variable).
- Change from baseline to 6 month follow-up Euro-Qol (EQ-5D) index (as a continuous variable).
- Modified American College of Rheumatology (ACR) ACR20, ACR50, ACR70.

Detailed definitions for the original analysis as well as all subsequent analyses will be included in respective statistical analysis plans (SAPs).

#### 9.4. Data Sources

The US Corrona RA Registry is the data source for this study. It is an independent, prospective, national, observational cohort. Patients are recruited from 187 private and academic sites across 43 states, with 799 providers participating. Providers and subjects complete study questionnaires approximately every 6 months at routine clinic encounters. As of September 2019, the Corrona database included information on 53,438 patients with RA. Data on 403,679 patient visits and 192,141 patient-years of follow-up observation time have been collected, with a mean patient follow-up of 4.48 (median 3.24) years. Data are collected on subjects for as long as they consent to remain in the study.

# 9.5. Study Size

Power calculations (below) indicate that to detect a reasonable difference of 15% in the percentage meeting MCID in CDAI, about 300-500 patients per group would be needed.

With the following assumptions:

- Consider the dichotomous outcome of meeting MCID in CDAI.
- We would like to have 90% power to detect a difference between the 2 groups in percentage meeting MCID in CDAI.
- We would like to have a low chance (alpha of 5%) of declaring that there is a difference in the outcomes between the 2 groups when in actuality there is not (type I error).

The following Table 1, gives the number needed per group and total number needed for different scenarios of meeting MCID for CDAI and percent of patients who are available under common support (eg, percent of patients in the control group that are similar enough to the treatment group so that we are comfortable that the 2 cohorts are similar). If we assume that the percentage meeting MCID in CDAI is 50%, the following sample sizes are required.

**Table 1.** Sample Size Determination

| Difference<br>between the 2<br>groups in<br>percentage<br>meeting MCID<br>in CDAI that can<br>be detected | Analyzable Data<br>Set, N per group | % under common support | N per group<br>required to<br>recruit | Total N<br>required to<br>recruit |
|---|---|---|---|---|
| 10% | 535 | 50% | 1070 | 2140 |
| 10% | 535 | 75% | 713 | 1426 |
| 15% | 237 | 50% | 474 | 948 |
| 15% | 237 | 75% | 316 | 632 |
| 20% | 131 | 50% | 262 | 524 |
| 20% | 131 | 75% | 175 | 350 |
| 25% | 84 | 50% | 168 | 336 |
| 25% | 84 | 75% | 112 | 224 |

Under different scenarios for projections of the total number of tofacitinib 11 mg QD initiators over time, it was estimated that there would be about 180-220 tofacitinib 11 mg QD initiators with 6 month follow-up visits by the end of 2018.

# 9.6. Data Management

Statistical analyses will be performed using Statistical Analysis System (SAS) Version 9.4 (SAS Institute, Cary, NC) and STATA Version 15 (StataCorp, LP, College Station, TX).

#### 9.7. Data Analysis

Patients initiating tofacitinib during or after February 2016 with a six-month follow-up visit (+/- 3 months) will be considered for analysis. Patient and disease characteristics at initiation for the two cohorts of 11 mg QD and 5 mg BID will be considered. Propensity score matching and adjustment for covariates will be used to identify a balanced, matched subset of patients to use in final analyses.

The primary outcome will be minimum clinically important difference (MCID) improvement as defined by difference in CDAI from initiation to 6 month visit (dichotomous variable). Secondary outcomes at the 6 month visit (follow-up): change in CDAI from initiation to follow-up, achievement of remission (CDAI\(\leq 2.8\)) and achievement of low disease activity (LDA) (CDAI\(\leq 10\)), achievement of improvement from baseline to follow-up in HAQ of 0.22 and change from baseline to 6 month follow-up HAQ, modified DAS, DAS ESR, DAS CRP, patient pain, patient fatigue, EQ5D index, modified ACR20/50/70. Sensitivity analysis, will be performed if needed.

Detailed methodology for the original analysis as well as all subsequent analyses is documented in respective SAPs, which are dated, filed and maintained by Pfizer. The SAP may modify the plans outlined in the protocol; any major modifications of primary endpoint definitions or their analyses would be reflected in a protocol amendment.

## 9.8. Quality Control

The Corrona registry has standard operating procedures in place to monitor, perform edit and logic checks, and make corrections to the data, as necessary. Specifically, the data for each site is reviewed by the Quality Department or other delegated Corrona representative for completeness and internal consistency at regular intervals. The Quality Department generates a list of queries for each site, sends to the clinical site coordinator, and requests verification or correction for each query within 14 days. The Quality Department or other designated Corrona representative enters corrected data onto the Corrona database. An audit trail of all corrections to the data, and the personnel making and date of corrections, is stored with the data in the Corrona database.

#### 9.9. Limitations of the Research Methods

This study has a number of limitations. Patient characteristics and access to medications can vary substantially between countries, due to payer and regulatory differences, thus these results may be less applicable outside of the US. Propensity score (PS) methods are intended to adjust for non-random treatment assignment, however, the possibility of bias and endpoint misclassification remains for observational studies. Furthermore, while we accounted for the most clinically significant variables, unmeasured residual confounding is a possibility.

# 9.10. Other Aspects

Not applicable.

#### 10. PROTECTION OF HUMAN SUBJECTS

#### 10.1. Patient Information

This study involves data that exist in anonymized structured format and contain no patient personal information.

#### 10.2. Patient Consent

As this study involves anonymized structured data, which according to applicable legal requirements do not contain data subject to privacy laws, obtaining informed consent from patients by Pfizer is not required.

## 10.3. Institutional Review Board (IRB)/Independent Ethics Committee (IEC)

IRB/IEC approvals/waivers not required.

# 10.4. Ethical Conduct of the Study

The study will be conducted in accordance with legal and regulatory requirements, as well as with scientific purpose, value and rigor and follow generally accepted research practices described in Guidelines for Good Pharmacoepidemiology Practices (GPP) issued by the International Society for Pharmacoepidemiology (ISPE), Good Epidemiological Practices (GEP) guidelines issued by the International Epidemiological Association (IEA).

# 11. MANAGEMENT AND REPORTING OF ADVERSE EVENTS/ADVERSE REACTIONS

This study involves data that exist as structured data by the time of study start.

In these data sources, individual patient data are not retrieved or validated, and it is not possible to link (ie, identify a potential association between) a particular product and medical event for any individual. Thus, the minimum criteria for reporting an adverse event (AE) (ie, identifiable patient, identifiable reporter, a suspect product, and event) cannot be met.

#### 12. PLANS FOR DISSEMINATING AND COMMUNICATING STUDY RESULTS

In the event of any prohibition or restriction imposed (eg, clinical hold) by an applicable competent authority in any area of the world, or if Corrona becomes aware of any new information which might influence the evaluation of the benefits and risks of a Pfizer product, Pfizer should be informed immediately.

The protocol will be disclosed at clinical trials.gov website along with the final study results. In addition, the study results will be submitted to national and international medical conferences and a final publication will be developed and submitted to an indexed, peer-reviewed medical journal in the area of rheumatology. Results from the interim/full analysis may also be reported to European Medicines Agency (EMA) to support MR submission.

#### 13. REFERENCES

- 1. Fleischmann R, Cutolo M, Genovese MC, et al. Phase IIb dose-ranging study of the oral JAK inhibitor tofacitinib (CP-690,550) or adalimumab monotherapy versus placebo in patients with active rheumatoid arthritis with an inadequate response to disease-modifying antirheumatic drugs. Arthritis Rheum 2012;64:617-29.
- 2. Kremer JM, Bloom BJ, Breedveld FC, et al. The safety and efficacy of a JAK inhibitor in patients with active rheumatoid arthritis: results of a double-blind, placebo-controlled phase IIa trial of three dosage levels of CP-690,550 versus placebo. Arthritis Rheum 2009;60:1895-905.
- 3. Kremer JM, Cohen S, Wilkinson BE, et al. A phase IIb dose-ranging study of the oral JAK inhibitor tofacitinib (CP-690,550) versus placebo in combination with background methotrexate in patients with active rheumatoid arthritis and an inadequate response to methotrexate alone. Arthritis Rheum 2012;64:970-81.
- 4. Tanaka Y, Suzuki M, Nakamura H, et al. Phase II study of tofacitinib (CP-690,550) combined with methotrexate in patients with rheumatoid arthritis and an inadequate response to methotrexate. Arthritis Care Res (Hoboken) 2011;63:1150-8.
- 5. Tanaka Y, Takeuchi T, Yamanaka H, et al. Efficacy and safety of tofacitinib as monotherapy in Japanese patients with active rheumatoid arthritis: a 12-week, randomized, phase 2 study. Mod Rheumatol 2015;25:514-21.
- 6. Burmester GR, Blanco R, Charles-Schoeman C, et al. Tofacitinib (CP-690,550) in combination with methotrexate in patients with active rheumatoid arthritis with an inadequate response to tumour necrosis factor inhibitors: a randomised Phase 3 trial. Lancet 2013;381:451-60.
- 7. Fleischmann R, Kremer J, Cush J, et al. Placebo-controlled trial of tofacitinib monotherapy in rheumatoid arthritis. N Engl J Med 2012;367:495-507.
- 8. Kremer J, Li Z-G, Hall S, et al. Tofacitinib in combination with nonbiologic disease-modifying antirheumatic drugs in patients with active rheumatoid arthritis: a randomized trial. Ann Intern Med 2013;159:253-61.
- 9. Lee EB, Fleischmann R, Hall S, et al. Tofacitinib versus methotrexate in rheumatoid arthritis. N Engl J Med 2014;370:2377-86.
- 10. van der Heijde D, Tanaka Y, Fleischmann R, et al. Tofacitinib (CP-690,550) in patients with rheumatoid arthritis receiving methotrexate: twelve-month data from a twenty-four-month phase III randomized radiographic study. Arthritis Rheum 2013;65:559-70.
- 11. van Vollenhoven RF, Fleischmann R, Cohen S, et al. Tofacitinib or adalimumab versus placebo in rheumatoid arthritis. N Engl J Med 2012;367:508-19.

- 12. Fleischmann R, Mysler E, Hall S, et al. Efficacy and safety of tofacitinib monotherapy, tofacitinib with methotrexate, and adalimumab with methotrexate in patients with rheumatoid arthritis (ORAL Strategy): a phase 3b/4, double-blind, head-to-head, randomised controlled trial. Lancet 2017;390:457-68.
- 13. Wollenhaupt J, Silverfield J, Lee EB, et al. Safety and efficacy of tofacitinib, an oral Janus kinase inhibitor, for the treatment of rheumatoid arthritis in open-label, longterm extension studies. J Rheumatol 2014;41:837-52.
- 14. Yamanaka H, Tanaka Y, Takeuchi T, et al. Tofacitinib, an oral Janus kinase inhibitor, as monotherapy or with background methotrexate, in Japanese patients with rheumatoid arthritis: an open-label, long-term extension study. Arthritis Res Ther 2016;18:34.
- 15. Wollenhaupt J, Lee EB, Curtis JR, et al. Safety and efficacy of tofacitinib for up to 9.5 years in the treatment of rheumatoid arthritis: final results of a global, open-label, long-term extension study. Arthritis Res Ther 2019;21:89.
- 16. Kremer JM. The Corrona US registry of rheumatic and autoimmune diseases. Clin Exp Rheumatol 2016;34:S96-S9.

#### 14. LIST OF TABLES

#### 15. LIST OF FIGURES

Not applicable.

#### ANNEX 1. LIST OF STAND ALONE DOCUMENTS

None.

## ANNEX 2. ENCEPP CHECKLIST FOR STUDY PROTOCOLS

Not applicable.

#### ANNEX 3. ADDITIONAL INFORMATION

Not applicable.